CLINICAL TRIAL: NCT05503589
Title: The Psychological Effect of the Covid-19 Pandemic on Turkish Intern Students
Brief Title: The Psychological Effect of the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Gamze Kurt, associate professor, Kutahya Health Sciences University
Other Study IDs: Covid-saliva
Record Dates: First submitted 2022-08-15; First posted 2022-08-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Psychological Distress
Keywords: psychological distress; Covid-19; saliva cortisol
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The unstimulated saliva samples of the participants were collected using the spitting method into the supplied polypropylene eppendorf tubes. Saliva samples collected in eppendorf tubes were centrifuged at 3,220 rpm for 10 minutes and stored at -20°C until the day of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- student group: have taken the professional practice/internship lecture and be practicing in the hospital
- control group: who routinely work during the pandemic

SUMMARY:
At the end of 2019, the novel coronavirus disease (Covid-19), which emerged in China, has become a public health emergency of international concern. Disease outbreaks both affect the physical and psychological health of individuals. The aim of this study was to investigate the levels of stress, anxiety, depression, and Covid-19 fear in health sciences intern students during the Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria for students:

* be over 18 years old
* have taken the professional practice/internship lecture
* be practicing in the hospital
* not have any disease

Inclusion Criteria for control:

* over the age of 18
* without any disease
* who routinely work during the pandemic

Exclusion Criteria:

* body mass index (BMI) <17 kg/m2
* any chronic illness, psychological disorder, and perception problem
* be dental operation or significant damage to the teeth or oral mucosa

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: intern students at the Faculty of Health Sciences of Kutahya Health Sciences University
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The Fear of Covid-19 Scale | 5 minutes
  The Fear of Covid-19 Scale (FCV-19S) is an assessment instrument developed to measure the fear levels of individuals due to Covid-19. The scale consists of seven items in a five-point Likert type. The total score is calculated by summing seven items score (ranging from 7-35). The high scale score indicates great fear of Covid-19.
Depression Anxiety and Stress Scale | 10 minutes
  Depression Anxiety and Stress Scale (DASS) is a self-report scale that evaluates depression, anxiety, and stress state over the past week. The scale consists of a total of 42 items, with 14 items in each of the depression, anxiety and stress dimensions. DASS items have a four-point Likert-type rating.The total scores each dimension of the scale range from 0 to 42. The high scores each of the depression, anxiety and stress dimensions indicate that the individual has a related problem.
Saliva cortisol level | 15 minutes
  The solid-phase sandwich ELISA (Enzyme Linked-Immuno-Sorbent Assay) method was used with immunoassay kits to measure the cortisol level.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze KURT, Ph.D., Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Sciences University- Health Sciences Faculty, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No